CLINICAL TRIAL: NCT06843226
Title: The Association Between Prior Exposure to Dengue Tetravalent Vaccine (Live, Attenuated) (TDV) and Dengue Hospitalization in a Pediatric and Adolescent Population: A Nested Case-Control Post-Authorization Effectiveness Study
Brief Title: A Study in Children and Adolescents on the Effectiveness of Takeda's Licensed Dengue Vaccine TDV Against Hospitalization Due to Dengue Disease
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: DEN-401; EUPAS1000000218 (Registry Identifier: EUPAS Number)
Record Dates: First submitted 2025-02-20; First posted 2025-02-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Dengue Fever
Keywords: Dengue Tetravalent Vaccine (Live, Attenuated) (TDV)
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Immunoglobulin G (IgG) enzyme-linked immunosorbent assay (ELISA) baseline testing for the cohort participants participating in the nested case control investigation and reverse transcription polymerase chain reaction (RT PCR) testing for clinically diagnosed dengue (CCD) hospitalised cohort participants to confirm virologically confirmed dengue (VCD).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nested Case-control Participants: The cohort will include case and control participants. Case participants who are hospitalized and meet the study inclusion and exclusion criteria for cases, have CDD, and have a confirmed positive RT-PCR test result (VCD) will be ascertained by active hospital surveillance.
  Control participants who are matched to a case and meet the study inclusion and exclusion criteria for controls but have not been hospitalized with VCD on or before their case's index date (first date of hospitalization for CDD for potential cases) will be interviewed.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The main aim of this study is to collect more information on the effectiveness of TDV when used in a pilot public vaccination program for children and adolescents participating in a community-based cohort in Southeast Asian countries where TDV is already approved for use.

The study will include cohort participants (individual follow-up of 3 years) who may or may not later be vaccinated with TDV as part of a pilot public vaccination program in the study countries. The study will investigate if cohort participants who were vaccinated with TDV have less hospital stays due to dengue than cohort participants who were not vaccinated with TDV. The study will also provide further information on the effectiveness of TDV against the least common dengue virus serotypes (DENV-3 and DENV-4).

ELIGIBILITY:
Inclusion Criteria:

Cohort:

To be eligible for inclusion in the study cohort, participants must meet the following inclusion criteria:

1. The participant is a child or adolescent eligible to be vaccinated with TDV as part of a vaccination program planned in the study area.
2. The participant's family do not intend to migrate away from the cohort hospital catchment area within 3 years of his/her enrollment into the study cohort.
3. The participant's parent or legally acceptable representative (LAR) signs and dates a written informed consent form (ICF), and any required privacy authorization where applicable, prior to the initiation of any study procedures, after the nature of the study has been explained according to local regulatory requirements.
4. The participant signs and dates an age-appropriate assent form prior to the initiation of any study procedures, after the nature of the study has been explained according to local regulatory requirements.
5. The participant's parent or LAR agrees that a baseline blood sample may be taken from the participant.

Cases:

To be eligible for inclusion as a case, participants must meet the following inclusion criteria:

1. The participant is part of the cohort.
2. The participant is hospitalized and clinically diagnosed with dengue.
3. The participant has a blood sample available that was taken preferably within 5 days of fever onset and/or onset of symptoms compatible with dengue.
4. The participant tested positive for dengue by RT-PCR.

Controls:

To be eligible for inclusion as a matched control, participants must meet the following inclusion criteria:

1. The participant is part of the cohort.
2. The participant had not been hospitalized with VCD at any point between enrollment in the cohort and the index date (that is, when his/her matched case was hospitalized with CDD).
3. The participant is a resident in the same neighbourhood as the matched case.
4. The participant's date of birth is in the same calendar year as the matched case.

Exclusion Criteria

Cases:

To be eligible for inclusion as a case participants must not meet any of the following criteria:

1. The participant has been vaccinated with TDV, a tetravalent, live attenuated, chimeric dengue vaccine in a yellow fever 17D backbone (CYD-TDV), or an investigational dengue vaccine prior to cohort enrollment.
2. Contraindications as per the locally approved label/product information leaflet.

Controls:

To be eligible for inclusion as a control participants must not meet any of the following criteria:

1. The participant has been vaccinated with TDV, CYD-TDV, or an investigational dengue vaccine prior to cohort enrollment.
2. Contraindications as per the locally approved label/product information leaflet.
3. The participant could not be contacted at the time of being selected as a control.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric and/or adolescent residents in the study area who are age-eligible for vaccination with TDV as part of a pilot public vaccination program.
Sampling Method: Non-Probability Sample
Enrollment: 70000 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospitalization Due to VCD of Any Dengue Serotype in Unvaccinated and Fully Vaccinated Participants | Up to Month 36
  Number of participants hospitalized due to VCD of any dengue serotype in unvaccinated and fully vaccinated participants.

SECONDARY OUTCOMES:
Hospitalization Due to VCD By Each Infecting Dengue Serotype (DENV-1, DENV-2, DENV-3, DENV-4) in Unvaccinated and Fully Vaccinated Participants | Up to Month 36
  Number of participants hospitalized due to VCD with each infecting dengue serotype (dengue virus [DENV]-1, DENV-2, DENV-3, and DENV-4) in unvaccinated and fully vaccinated participants will be reported.
Hospitalization Due to VCD by Baseline Dengue Serostatus (Seronegative and Seropositive) of Any Dengue Serotype in Unvaccinated and Fully Vaccinated Participants | Up to Month 36
  Number of participants hospitalized due to VCD with dengue serostatus (seronegative and seropositive) of any dengue serotype in unvaccinated and fully vaccinated participants will be reported.
Hospitalization Due to VCD By Each Infecting Dengue Serotype and Baseline Dengue Serostatus in Unvaccinated and Fully Vaccinated Participants | Up to Month 36
  Number of participants hospitalized due to VCD by each infecting dengue serotype and baseline dengue serostatus (DENV-1 in baseline seronegative, DENV-2 in baseline seronegative, DENV-3 in baseline seronegative, DENV-4 in baseline seronegative, DENV-1 in baseline seropositive, DENV-2 in baseline seropositive, DENV-3 in baseline seropositive, and DENV-4 in baseline seropositive) in unvaccinated and fully vaccinated participants will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- Thailand (3):
  - Pattaya Patamakhun Hospital, Bang Lamung, Changwat Chon Buri
  - Nakhon Phanom hospital, Nakhon Phanom, Changwat Nakhon Phanom
  - Phra Nakhon Si Ayutthaya Hospital, Mueang Phra Nakhon Si Ayutthaya, Phra Nakhon Si Ayutthaya

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/2aae75732b0e49cd??page=1&idFilter=DEN-401